CLINICAL TRIAL: NCT02413827
Title: A Phase 1 Safety Pilot/Phase II, Open-label Study of Varlilumab (CDX-1127) in Combination With Ipilimumab and CDX-1401 in Patients With Unresectable Stage III or Stage IV Melanoma
Brief Title: A Study of Varlilumab (Anti-CD27) and Ipilimumab and CDX-1401 in Patients With Unresectable Stage III or IV Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Feasibility concerns due to changes in standard of care
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX1127-03
Record Dates: First submitted 2015-03-25; First posted 2015-04-10 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Unresectable Stage III or Stage IV Melanoma
Keywords: Yervoy™, CDX-1401
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase l: varlilumab and ipilimumab (Experimental)
  Interventions: Drug: Combination of varlilumab and ipilimumab
- Phase ll: varlilumab & ipilimumab, +/- CDX-1401 & poly-ICLC. (Experimental)
  Interventions: Drug: Cohort A: varlilumab & ipilimumab; Cohort B: varlilumab, ipilimumab, CDX-1401 & poly-ICLC

INTERVENTIONS:
Drug: Combination of varlilumab and ipilimumab — Eligible patients will receive assigned treatments once every 3 weeks for a total of 4 treatments.
  Phase l dose: The planned dose of varlilumab will be dependent on the cohort assigned at enrollment. Varlilumab doses are 0.3 mg/kg or 3 mg/kg. Ipilimumab dose is 3 mg/kg.
  Arms: Phase l: varlilumab and ipilimumab
Drug: Cohort A: varlilumab & ipilimumab; Cohort B: varlilumab, ipilimumab, CDX-1401 & poly-ICLC — Eligible patients will receive assigned treatments once every 3 weeks for a total of 4 treatments.
  Phase ll dose: The planned dose of varlilumab will be established from Phase I. Ipilimumab dose is 3 mg/kg. Patients assigned to receive CDX-1401 will receive a dose of 1 mg along with 2 mg poly-ICLC.
  Arms: Phase ll: varlilumab & ipilimumab, +/- CDX-1401 & poly-ICLC.

SUMMARY:
This is a study to determine the clinical benefit (how well the drug works), safety and tolerability of combining a) varlilumab and ipilimumab and b) varlilumab, ipilimumab, CDX-1401 and poly-ICLC. The study will enroll patients with unresectable Stage III or Stage IV melanoma.

DETAILED DESCRIPTION:
Varlilumab is a fully human monoclonal antibody that binds to a molecule called CD27 found on certain immune cells and may act to promote anti-tumor effects.

Yervoy™ (Ipilimumab) is a human monoclonal antibody that blocks CTLA-4, a protein receptor that downregulates the immune system.

CDX-1401 is a vaccine made of a fully human monoclonal antibody linked to NY-ESO-1 and is designed to deliver NY-ESO-1 to professional antigen presenting cells for generating robust immune responses against cancer cells expressing NY-ESO-1. CDX-1401 is administered with poly-ICLC, an adjuvant that enhances vaccine-induced immune responses.

This study will evaluate the safety, tolerability and efficacy of varlilumab and ipilimumab, with or without the addition of CDX-1401/poly-ICLC, in patients with melanoma.

Eligible patients that enroll in the Phase I portion of the study will be assigned to one of two possible dose levels of varlilumab in combination with 3 mg/kg ipilimumab. The first phase of the study will test the safety profile of the combination and determine which dose of varlilumab will be studied in Phase II of the study.

During Phase II, up to 48 patients whose tumors do not express NY-ESO-1, will receive the recommended dose of varlilumab determined from Phase I with 3 mg/kg ipilimumab. Up to 24 patients whose tumors express NY-ESO-1 will receive the recommended dose of varlilumab combined with 3 mg/kg ipilimumab and 1 mg CDX-1401 along with 2 mg poly-ICLC.

All patients enrolled in the study will be closely monitored to determine if there is a response to the treatment as well as for any side effects that may occur.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologic diagnosis of melanoma.
2. Unresectable Stage III or IV disease
3. Documented progressive disease based on radiographic, clinical or pathologic assessment.
4. No more than three prior anticancer regimens (BRAF/MEK inhibitors, IL-2 or investigational agents) including no more than one chemotherapy-containing regimen for advanced (recurrent, locally advanced or metastic) disease.
5. Measurable disease.
6. Life expectancy ≥ 12 weeks.
7. If of childbearing potential (male or female), agrees to practice an effective form of contraception during study treatment and for at least 70 days following last treatment.
8. Availability of tumor tissue for central laboratory analyses.

Key Exclusion Criteria:

1. Previous treatment with anti-CD27 antibody, ipilimumab or other anti-CTLA-4 targeted therapies. Previous therapy with other checkpoint blockers such as anti-PD-1 or anti-PD-L1 is acceptable, unless treatment was discontinued for intolerance.
2. For patients enrolled to Phase II Cohort B: Previous administration of vaccine therapy targeting NY-ESO-1.
3. BRAF/MEK inhibitors within 2 weeks prior to first dose of study treatment.
4. Chemotherapy within 21 days or at least 5 half-lives (whichever is shorter) prior to first dose of study treatment.
5. Monoclonal based therapies within 4 weeks and all other immunotherapy within 2 weeks prior to first dose of study treatment.
6. Systemic radiation therapy within 4 weeks, focal radiotherapy within 2 weeks and radiopharmaceuticals (strontium, samarium) within 8 weeks prior to first dose of study treatment.
7. Ocular Melanoma
8. Other prior malignancy, except for adequately treated basal or squamous cell skin cancer or in situ cancers; or any other cancer from which the patient has been disease-free for at least 3 years.
9. Active, untreated central nervous system metastases.
10. Active autoimmune disease or documented history of autoimmune disease.
11. Active diverticulitis
12. Significant cardiovascular disease including CHF or poorly controlled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-11-02 (Actual); Study Completion 2016-11-09 (Actual)

PRIMARY OUTCOMES:
Phase l: Safety and tolerability of varlilumab in combination with ipilimumab as measured by incidences of drug related adverse events (AEs), serious drug related AEs, dose-limiting toxicities and laboratory test abnormalities. | Safety follow-up is 70 days from last study drug dose.
Phase ll: The objective response rate (ORR) is defined as the proportion of patients who achieve radiographic partial or complete response (PR or CR) according to the mWHO tumor response criteria. | Up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - California Pacific Medical Center Research Institute, San Francisco, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - University of Colorado, Aurora, Colorado
  - Georgetown University School of Medicine, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology Sarah Cannon Research Institute, Nashville, Tennessee